CLINICAL TRIAL: NCT00012246
Title: A Trial Of Vaccination With The Carcinoembryonic Antigen (CEA) Peptide Cap 1-6D With Montanide ISA 51 Adjuvant Or Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) In HLA-A2+ Patients With CEA Producing Adenocarcinomas Of Gastrointestinal (GI) Tract Origin
Brief Title: Vaccine Therapy in Treating Patients With Cancer of the Gastrointestinal Tract
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively Terminated
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068497; UTMB-00-297; NCI-931
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastric Cancer; Pancreatic Cancer; Small Intestine Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; small intestine adenocarcinoma; localized gallbladder cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; localized extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; adenocarcinoma of the esophagus; adenocarcinoma of the colon; adenocarcinoma of the rectum; adenocarcinoma of the gallbladder; adenocarcinoma of the extrahepatic bile duct; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Adenocarcinoma Of Esophagus | interventions — incomplete Freund's adjuvant; sargramostim

INTERVENTIONS:
Biological: carcinoembryonic antigen peptide 1-6D
Biological: incomplete Freund's adjuvant
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of two different vaccines in treating patients who have cancer of the gastrointestinal tract.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether immunization with carcinoembryonic antigen (CEA) peptide 1-6D (CAP 1-6D) emulsified in Montanide ISA-51 adjuvant or dissolved in sargramostim (GM-CSF) can generate CAP 1-6D-specific T cells in patients with CEA-producing adenocarcinomas of gastrointestinal tract origin.
* Determine whether vaccination with CAP 1-6D can generate cytotoxic T cells against CEA-expressing tumors in these patients.
* Determine whether this vaccine can produce antitumor responses in these patients.
* Determine the frequency and severity of toxic effects associated with this vaccine in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive carcinoembryonic antigen peptide 1-6D (CAP 1-6D) emulsified in Montanide ISA-51 adjuvant subcutaneously on day 1.
* Arm II: Patients receive CAP 1-6D dissolved in sargramostim (GM-CSF) intradermally on day 1.

Treatment repeats in both arms every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 weeks and then as necessary.

PROJECTED ACCRUAL: A total of 10-36 patients (5-18 per arm) will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II, III, or IV adenocarcinoma of the gastrointestinal tract originating in 1 of the following:

  * Esophagus
  * Stomach
  * Pancreas
  * Small intestine
  * Colon or rectum
  * Gall bladder
  * Extrahepatic bile ducts
  * Ampulla of Vater
* Completed standard therapy and at risk of recurrent disease OR has relatively stable metastatic disease and a life expectancy of at least 6 months
* Carcinoembryonic antigen (CEA)-producing tumor as evidenced by detectable blood levels of CEA or positive for CEA on immunohistochemical staining
* Human Leukocyte Antigen (HLA)-A2+

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Southwest Oncology Group (SWOG) 0-1

Life expectancy:

* See Disease Characteristics

Hematopoietic:

* White Blood Count (WBC) at least 4,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Serum Glutamic Oxalacetic Transaminase (SGOT) or Serum Glutamic Pyruvic Transaminase (SGPT) no greater than 3 times upper limit of normal
* Hepatitis B and C negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No other prior malignancy unless currently disease free and off all therapy for that malignancy

  * Early skin cancer allowed
* No AIDS
* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 30 days after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* At least 4 weeks since prior surgery

Other:

* No other concurrent therapy for malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Production of CAP 1-6D T cells
Production of cytotoxic T cells
Antitumor response
Frequency and severity of toxic effects

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Whitehead, MD, Study Chair — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States